CLINICAL TRIAL: NCT06100211
Title: A Prospective Observational Study of the Impact on the Gut Microbiome in HIV-infected Individuals in Manchester, UK, When Switching From One Class of Antiretroviral Drugs or Delivery Method to Another Class or Delivery Method.
Brief Title: HIV and Changes in the Gut Microbiome After Changes in Antiretroviral Therapy (ART)
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Gabriella Lindergard, Clinical Lecturer in Nursing, University of Manchester
Other Study IDs: 333914
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
Keywords: HIV; Gut microbiome; Antiretroviral drugs
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART switch group: These are individuals who complete a planned switch of ART regimen from one class of drugs or delivery method to another.
- Control group: This group continue on their stable ART regimen.

SUMMARY:
This is a study that aims to contribute to the understanding of how antiretroviral therapy effects the gut microbiome which, if known, could inform decisions about drug choices at an individual level.

The gut health is extremely important for all aspects of a persons wellbeing both at the level of the body and the brain. In recent years there has been much interest and better understanding of the role of the bacteria, viruses and other microorganisms that live in the human gut (the gut microbiome). It is known that disturbing the balance between the different species of bacteria in the gut can have consequences including diarrhoea, inflammatory and autoimmune conditions and has also been linked to obesity.

There are big differences in the gut microbiome composition seen in people with untreated HIV infection compared with non-infected individuals. This disrupted balance does not seem to be restored when starting on antiretroviral therapy. Different classes of antiretrovirals seem to have different effects but this has been hard to establish because studies aiming to look at this has been large population studies where it can be hard to tease out cause and effect.

In this study the investigators are instead aiming to compare an individual with themselves by comparing the bacterial gut microbiome before the person switches from one class of antiretroviral treatment to another or switches the delivery method of that drug, with the bacterial gut microbiome 3-8 weeks after the switch.

The investigators hope that if this can be understood the effects different classes and delivery methods of antiretroviral have on an individual's gut microbiome, can be taken into account when deciding on the best HIV therapy for a person. In the long term, this would lessen the negative effects of being on a life-long treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Willing to undergo stool sample collection on two occasions.
* Able to give written, informed consent.
* Have evidence of HIV infection
* Have been on stable antiretroviral treatment for the previous ≥12months.
* Planning to switch ART regimen from one class of drugs or delivery method to another.

Exclusion Criteria:

* HIV viral load >50 copies/ml blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected individuals on stable antiretroviral treatment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
To measure changes in diversity and abundance of bacterial species in stool sample collected before and after a change of ART. | 3-8 weeks
  The number of different bacterial species and the abundance of these species will be measured by shallow shotgun sequencing before and after the change in antiretroviral treatment.

SECONDARY OUTCOMES:
To link level of bacterial diversity with different ART regiments. | 3-8 weeks
  To measure the level of change in the number and the abundance of bacterial species after a change of antiretroviral treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No